CLINICAL TRIAL: NCT00638404
Title: Predicting Severity of Postoperative Pain After Surgery
Brief Title: Severity Postoperative Pain Prediction
Status: Terminated | Type: Observational
Why Stopped: Further evaluation determined it was not feasible to enroll the post-partum tubal ligation group at our facility
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Other Study IDs: Pain Prediction
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Results first posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2017-08

CONDITIONS: Anxiety; Pain; Postoperative Pain
Keywords: Preoperative somatic questions; Preoperative audio tone evaluations; Preoperative anxiety and previous experience with postop pain
MeSH Terms: conditions — Anxiety Disorders; Pain; Pain, Postoperative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Elective Cesarean Sections-this portion completed
- 3: Any in-patient gynecologic procedure- this portion completed

SUMMARY:
A simple preoperative evaluation assessing level of anxiety, anticipated pain, and intensity rating of audio tone will predict the severity of postoperative pain after surgery.

DETAILED DESCRIPTION:
The purpose of this study would be to determine the predictive value of a simple to perform preoperative evaluation in assessing level of anxiety, anticipated pain and the intensity rating of an audio tone to predict level of postoperative pain after surgery.

Study Design: A total of 400 evaluable patients will be studied using the various surgical populations listed. For statistical purposes, the following will be the surgical population by procedure. Two hundred healthy ASA I-II women scheduled for elective cesarean section, one hundred scheduled for elective postpartum tubal ligations, and one hundred scheduled for elective inpatient gynecological surgeries (such as total vaginal hysterectomy, total abdominal hysterectomy) will be consented and enrolled in the study. Normal baseline vital signs will be obtained and recorded as part of usual preoperative assessment for these patients. The patients will be asked about their current level of pain and to rate the intensity of a series of audio tones. At 18-24 hours postoperatively, and again at 36-48 hours postoperatively if applicable, research personnel will evaluate the severity of postoperative pain the patient has at rest and with movement (from supine to sitting upright), using a sliding pain scale from 0 to 100 mm, with 0 being no pain and 100 being the worst pain ever. Information on drug administered in the preoperative, intraoperative and postoperative period will be collected and recorded. The subject can also choose to allow us to follow-up with them in the future to evaluate current residual postoperative pain levels as needed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy ASA physical status class 1 or 2
* Aged 18 years or above
* Pregnant with intrauterine pregnancy of at least 36 weeks for cesarean sections

Exclusion Criteria:

* ASA >3
* < 36 weeks for Cesarean Section
* < 18 years of age

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: scheduled for elective cesarean section, non-pregnant subjects scheduled for inpatient gynecological surgeries
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2007-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter H. Pan, MSEE, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Forsyth Medical Center, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 200 Elective cesarean sections and 100 gynecological patients were enrolled prior to their surgery with presurgical testing completed. All subjects were then also seen postoperatively for followup
Pre-assignment Details: no randomization, only observational study
Groups:
- 1-elective Cesarean Section: Elective Cesarean Sections-preoperative questionnaire as well as audio testing completed prior to surgery with followup done 24 hours postoperatively
- 3-inpatient Gynecologic Procedures: Any in-patient gynecologic procedure-preoperative questionnaire as well as audio testing completed prior to surgery with followup done 24 hours postoperatively
Period: Overall Study
Arm/Group | 1-elective Cesarean Section | 3-inpatient Gynecologic Procedures
Started | 200 | 100
Completed | 192 | 100
Not Completed | 8 | 0
Not completed — Physician Decision | 8 | 0

BASELINE CHARACTERISTICS:
Groups:
- 1-elective Cesarean Sections: Elective Cesarean Sections-this portion completed
- 3-inpatient Gynecologic Procedures: Any in-patient gynecologic procedure- this portion completed
- Total: Total of all reporting groups
Arm/Group | 1-elective Cesarean Sections | 3-inpatient Gynecologic Procedures | Total
Number analyzed (Participants) | 192 | 100 | 292
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 192 | 100 | 292
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (4.8) | 44.5 (9.0) | 34.95 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 192 | 100 | 292
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 44 | 18 | 62
  Hispanic | 8 | 2 | 10
  White | 140 | 80 | 220
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 192 | 100 | 292

OUTCOME MEASURES:

1. Primary Outcome: Evoked Pain at 24 Hours VAS
Description: Outcome measure 0-100 Visual analog scale at 24 hours postoperatively, VAS of 0= no pain up to 100 =most severe pain
Time Frame: evoked pain at 24 hours
Population: evoked pain outcome-measured on a scale of 0=no pain up to 100=most severe pain imaginable.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 1-elective Cesarean Section: Elective Cesarean Sections-evoked pain score at 24 hours postoperative 0-100mmVAS
- 3-inpatient Gynecologic Procedures: Any in-patient gynecologic procedure-
Arm/Group | 1-elective Cesarean Section | 3-inpatient Gynecologic Procedures
Number analyzed (Participants) | 192 | 100
units on a scale | 44 (26) | 49.3 (30.7)
Statistical Analysis 1: Comparison: 1-elective Cesarean Section; Test type: Other — correlation of anxiety, anticipated pain medication use and anticipated pain to 24 hour evoked pain measured; p < .001, Spearman Correlation; anxiety to evoked pain is 0.24 (P<.001); anticipated pain to evoked pain is 0.33 (P<.001); anticipated pain medication to evoked pain is 0.33(P<.001)
Statistical Analysis 2: Comparison: 1-elective Cesarean Section; Test type: Other — correlation of anxiety to evoked pain at 24 hour; p < .001, Spearman Correlation
Statistical Analysis 3: Comparison: 1-elective Cesarean Section; Test type: Other — correlation of anticipated pain medication 24 hour evoked pain measured; p < .001, Spearman Correlation
Statistical Analysis 4: Comparison: 1-elective Cesarean Section; Test type: Other — correlation of anticipated pain to 24 hour evoked pain measured; p < .001, Spearman Correlation

2. Secondary Outcome: Anticipated Pain Medication Requirement
Description: measured on a scale of 0-5, with 0=no anticipated pain medication needed up to 5 =most anticipated pain medication required
Time Frame: 24 hours
Measure: Median (Full Range); unit: units on a scale
Groups:
- 1-elective Cesarean Section: Elective Cesarean Sections-anticipated pain medication required postoperative evaluated during preoperative evaluation
Arm/Group | 1-elective Cesarean Section | 3-inpatient Gynecologic Procedures
Number analyzed (Participants) | 192 | 100
units on a scale | 3 [0 to 5] | 3 [0 to 5]
Statistical Analysis 1: Comparison: 1-elective Cesarean Section; preoperative questionnaire evaluating anticipated amount of pain medication potentially needed postoperatively; 0= none at all up to 100=as much as possible; Test type: Other; p < .001, Spearman Correlation

3. Secondary Outcome: Anticipated Postoperative Pain at Preoperative Evaluation
Description: anticipated postoperative pain on a scale of 0-100mm with 0=no anticipated pain at all up to 100= worst anticipated pain imaginable
Time Frame: anticipated postoperative pain
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 1-elective Cesarean Section: Elective Cesarean Sections-anticipated pain postoperative obtained during preoperative evaluation
Arm/Group | 1-elective Cesarean Section | 3-inpatient Gynecologic Procedures
Number analyzed (Participants) | 192 | 100
units on a scale | 57 (26) | 60.8 (27.2)
Statistical Analysis 1: Comparison: 1-elective Cesarean Section; Test type: Other; p < .001, Spearman Correlation

4. Secondary Outcome: Anxiety
Description: measure of anticipated anxiety for on a scale of 0-100, with 0= not anxious at all up to 100 = most anxious
Time Frame: anticipated anxiety prior to surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 1-elective Cesarean Section: Elective Cesarean Sections preoperatively anxiety level
- 3-inpatient Gynecologic Procedures: Any in-patient gynecologic procedure-preoperative anxiety level on a scale of 0-not anxious at all up to 100=most anxious
Arm/Group | 1-elective Cesarean Section | 3-inpatient Gynecologic Procedures
Number analyzed (Participants) | 192 | 100
units on a scale | 52 (32) | 57.5 (34.8)
Statistical Analysis 1: Comparison: 1-elective Cesarean Section; Test type: Other — Correlation of; p < .001, Spearman Correlation

ADVERSE EVENTS:
Arm/Group | 1-elective Cesarean Sections | 3-inpatient Gynecologic Procedures
All-Cause Mortality (participants affected / at risk) | 0/192 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/192 | 0/100
Other Adverse Events (participants affected / at risk) | 0/192 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes